CLINICAL TRIAL: NCT04608253
Title: A Retrospective Analysis of the Diagnostic Performance of 11C-choline PET/CT for Detection of Hyperfunctioning Parathyroid Glands After Prior Negative or Discordant Imaging in Primary Hyperparathyroidism
Brief Title: A Retrospective Analysis of the Diagnostic Performance of 11C-choline PET/CT in Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/658
Record Dates: First submitted 2020-10-27; First posted 2020-10-29 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Primary Hyperparathyroidism; Primary Hyperparathyroidism Due to Adenoma
MeSH Terms: conditions — Hyperparathyroidism, Primary; Parathyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All enrolled subjects received an 11C-choline PET/CT prior to enrollment.: Patients with biochemically proven primary hyperparathyroidism who underwent parathyroid surgery after localization by means of 11C-choline PET/CT and negative or discordant first-line imaging
  Interventions: Diagnostic Test: 11C-choline PET/CT

INTERVENTIONS:
Diagnostic Test: 11C-choline PET/CT — 11C-choline PET/CT

SUMMARY:
The leading cause of primary hyperparathyroidism (pHPT) is a solitary adenoma (89%). The treatment of pHPT is generally surgical removal of the overactive parathyroid gland(s). Since a solitary adenoma is the predominant cause, parathyroid surgery is preferably performed through a minimally invasive parathyroidectomy (MIP) in which only the suspected adenoma causing the pHPT is resected in a focused manner. To facilitate the performance of a MIP, accurate preoperative imaging is pivotal. This study aimed to analyze the diagnostic performance of 11C-choline PET/CT after prior negative or discordant first-line imaging in patients with pHPT undergoing parathyroid surgery with an optimized imaging protocol.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion were ≥18 years old, diagnosed with biochemically confirmed pHPT, underwent a MIBI-SPECT/CT and/or cUS with negative or discordant results, and underwent a 11C-choline PET/CT followed by parathyroidectomy.

Exclusion Criteria:

Patients were excluded if they were known to have a germline mutation predisposing for familial hypocalciuric hypercalcemia (FHH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective single-center cohort study of patients with biochemically proven pHPT who underwent parathyroid surgery after localization by means of 11C-choline PET/CT and negative or discordant first-line imaging in a teaching and tertiary referral hospital in the Netherlands between 2015 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 11C-choline PET/CT | Until 6 months after parathyroid surgery
  Per-lesion sensitivity of 11C-choline PET/CT for the detection of overactive parathyroid glands
Positive predictive value of 11C-choline PET/CT | Until 6 months after parathyroid surgery
  Per-lesion positive predictive value of 11C-choline PET/CT for the detection of overactive parathyroid glands
Accuracy of 11C-choline PET/CT | Until 6 months after parathyroid surgery
  Per-lesion accuracy of 11C-choline PET/CT for the detection of overactive parathyroid glands

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Brouwers, MD PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request via the principle investigator